CLINICAL TRIAL: NCT05522907
Title: Comparative Study of Tumor Microenvironment Between Early and Advanced Prostate Cancer Through Multi-omics
Brief Title: Investigation of Tumor Microenvironment After CRPC Along With Before and After Neoadjuvant Therapy for Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021CRF-002
Record Dates: First submitted 2022-08-16; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
Keywords: Neoadjuvant; CRPC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From the beginning of the project for the past five years to the next three years, biospecimens from patients who received neoadjuvant therapy and underwent prostate cancer biopsy and underwent radical prostatectomy after 3-6 months of neoadjuvant therapy in the First Affiliated Hospital of Xi'an Jiaotong University.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant: From the beginning of the project for the past five years to the next three years, underwent prostate cancer biopsies at the First Affiliated Hospital of Xi'an Jiaotong University before neoadjuvant therapy, and underwent radical prostatectomy after 3-6 months of neoadjuvant therapy.
- CRPC: Patients with CRPC-diagnosed prostate cancer after initial continuous ADT therapy, with serum testosterone reaching castration levels (<50ng/dl or <1.7nmol/L) but with progressive disease, and who were diagnosed with CRPC at Xi'an Jiaotong University The First Affiliated Hospital did a prostate cancer biopsy.

SUMMARY:
In recent years, the clinical research of immunotherapy including PD-1 antibody and CD3 bispecific antibody in prostate cancer has been increasing day by day. The comparison with the analysis results of cancer tissues of advanced patients has important guiding significance for the application of these new treatment methods.

In a retrospective study, investigators plan to perform multi-omics analysis (including whole exome, RNAseq), immune cell characterization, and biopsy samples from prostate cancer primary biopsy, ADT neoadjuvant, and CRPC biopsy samples in the biobank. Protein and prostate cancer-specific antigen expression were analyzed by immunohistochemistry. The following questions are answered by comparing samples from different treatment stages in early and advanced stages: 1. Whether the immune environment becomes "cold" in the advanced stage; 2. Which immune cell populations have changed significantly; 3. Is the inhibitory immune microenvironment related to genes Mutations or suppressive immune cell populations.

DETAILED DESCRIPTION:
Prostate cancer is a high incidence of cancer in Europe and the United States. In recent years, due to factors such as increasing awareness of testing and an aging population, the incidence of prostate cancer in China has been increasing year by year, and it has become the sixth most common cancer in men. Most of the patients with middle-advanced prostate cancer respond to ADT treatment, but the vast majority of patients eventually develop castration-resistant prostate cancer (CRPC) after the disease recurs or continues to progress after castration treatment. The related drug resistance mechanism is mainly caused by abnormal AR signaling pathway, including AR gene amplification, AR splicing variant and AR coregulator activation and other factors. In recent years, studies have shown that inhibitory immune cell infiltration and immune microenvironment also promote the emergence of CRPC. The cytokine IL-23 secreted by infiltrating myeloid-derived suppressor cells (MDSCs) can activate the STAT3-RORγ pathway, which in turn activates the AR pathway, resulting in resistance to ADT and other AR-targeted therapies. In addition, advanced prostate cancer tissue has always been considered to be a relatively "cold" immune microenvironment with relatively little immune cell infiltration. Metastatic castration-resistant prostate cancer (mCRPC) lacks efficacy against immune checkpoint inhibitors such as PD-1, and only those with mismatch repair gene deficiency (dMMR) or microsatellite instability-high (MSI-H) have must benefit. Most studies have only focused on patients with advanced CRPC without systematically comparing the immune microenvironment of patients with early and advanced prostate cancer. Advances in next-generation sequencing (NGS) technologies have led to a greater understanding of genomic alterations in prostate cancer. The most common genomic abnormalities in this malignancy are the TMPRSS2-ETS transcription factor fusion, and mutations in TP53, AR, RB1, and PTEN/PIK3CA. Some of these abnormalities are already targeted with clinically available drugs. At present, there have been large-scale foreign research on prostate cancer, such as "The Cancer Genome Atlas" (TCGA), "International Cancer Genome Consortium" (ICGC), etc., and a western cancer omics research system has been established. In the Chinese Prostate Cancer Genome and Epigenome Atlas (CPGEA) study, the incidence of the hallmark ETS fusion (53% TCGA) was much lower in the Chinese prostate cancer population (9% CPGEA) in contrast to Western prostate cancer . Among Chinese prostate cancers, the highest gene fusion rates were SCHLAP1-UBE2E3 (29%) and PAOX-MTG1 (10%), and the researchers found that FOXA1 was the gene with the highest mutation rate (41%) in our Chinese prostate cancer patients. In terms of methylation, the Chinese cohort study is similar to the Western cohort, the prostate cancer genome is hypomethylated relative to normal prostate tissue, and the 5' untranslated region (UTR) and CpG island (CGI) are relatively hypermethylated, while the penetrance Introns, introns and repeat elements are hypomethylated. Megabase-scale partially methylated domains (PMDs) are widespread and affect up to half of the cancer genome, suggesting that tumor progression correlates with the extent of genome-wide hypomethylation.

Given the many differences in the genomes of Chinese and western prostate cancer patients, the response of Chinese prostate cancer patients to various treatments and the changes in gene, transcription, and translation levels after treatment may also be different from foreign prostate cancer patients. However, NGS data for Chinese prostate cancer patients before and after chemotherapy, endocrine therapy, radiotherapy, or immunotherapy are still missing. The NGS data of these patients before and after treatment will provide new drug design targets and new drug development ideas for prostate cancer treatment in China, and will also provide a solid theoretical basis for the optimization of existing treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* The patient was diagnosed with prostate cancer.
* The patient underwent neoadjuvant therapy or was diagnosed with CRPC.

Exclusion Criteria:

* When it is detected that the patient has a viral infection that interferes with the human genome, such as HIV infection, etc.
* Biopsy and/or surgically removed prostate cancer tissue was not eligible for the study.

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients who underwent prostate cancer biopsy before neoadjuvant therapy, underwent radical prostatectomy 3-6 months after neoadjuvant therapy.
  Patients were diagnosed with CRPC.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FFPE samples requirements | From the date of participants recruitment to the date of collection of at least 80 eligible FFPE samples, assessed up to 36 months.
  1. H&E stained slide (tumor area marked, tumor content >= 20%).
  2. Standard sample request:5-10 unstained slides, thickness 4-5um,0.6mm3 (matched to H&E slide).
Quality requirements for RNA extracted from FFPE samples | From the date of participants recruitment to the date of collection of at least 80 eligible FFPE samples, assessed up to 36 months.
  Standard sample request: more than 300ng total RNA, concentration: more than 20ng/ul, volume: more than 10 ul, DV200: more than 30%. Minimum sample request: more than 150ng total RNA, concentration: more than 20ng/ul, volume: more than 10 ul,DV200: more than 30%.
Quality requirements for DNA extracted from FFPE samples | From the date of participants recruitment to the date of collection of at least 80 eligible FFPE samples, assessed up to 36 months.
  Standard sample request: more than 2.2ug total RNA,concentration: more than 50ng/ul,volume: more than 10 ul,RIN: more than 8.Minimum sample request: more than 1.1ug total RNA,concentration: more than 50ng/ul,volume: more than 10 ul,RIN: more than 8.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, PhD, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China